CLINICAL TRIAL: NCT03656601
Title: Correlation Between Tridimensional Pelvic Floor Ultrasound and Quality of Life Scores Questionnaires in Nulliparous or Parous Women
Brief Title: Tridimensional Pelvic Floor Ultrasound and Quality of Life Scores Questionnaires in Nulliparous or Parous Women
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Maria Homem de Mello Bianchi, PhD of Gynecology Department, Federal University of São Paulo
Other Study IDs: 66574316.4.0000.5505
Record Dates: First submitted 2017-12-24; First posted 2018-09-04 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Urinary Incontinence; Anal Incontinence; Sexual Dysfunction; Self Esteem; Delivery
Keywords: 3D ultrasound; pelvic floor; delivery; quality of life
MeSH Terms: conditions — Urinary Incontinence; Encopresis; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vaginal delivery: Women that had only vaginal delivery
  Interventions: Diagnostic Test: 3D pelvic ultrasound
- Cesarean-section: Women that had only cesarean-section
  Interventions: Diagnostic Test: 3D pelvic ultrasound
- Nulliparous: Women without delivery
  Interventions: Diagnostic Test: 3D pelvic ultrasound

INTERVENTIONS:
Diagnostic Test: 3D pelvic ultrasound — 3D pelvic ultrasound by transperineal route

SUMMARY:
Evaluation of the impact of the delivery in the system of suspension and sustentation of pelvic floor, by 3D ultrasound and quality of life questionnaires.nt

DETAILED DESCRIPTION:
The pelvic floor is a complex group of muscle, fascia and connective tissue that recover the basis of the pelvic bones, forming the system of suspension and sustentation of the pelvic organs. Different events that happen during the life of women, like pregnancy, delivery, gain of weight and hormonal alterations from the menopause, may affects the strength of the muscles and of other structures that supports pelvic organs. The importance of the balance of the pelvic organs in maintenance of quality of life have been recognized in literature last years. Different studies established association between sexual disfunction and emotional dissatisfaction, as well as reduction of well-being in that women. The urinary incontinence and anal incontinence are also important factors that compromised quality of life and can provoke harmful effects over the self-esteem of women and diminish relationship. The 3D ultrasound (3D UD) is a non-invasive method, reproductible, and technically easy of evaluate the pelvic floor. Different routes may be used, but the transperineal is the most common. By this route is possible to evaluate the pelvic floor anatomy, as well as its disfunction into deep planes, what we can not afford only with the physical exam.

The objective was to evaluate the impact of the delivery on the pelvic floor, by the 3D ultrasound evaluation and to correlate it with the scores of sexual questionnaire (FSFI), urinary questionnaire (King´s) and anal incontinence questionnaire ( specific questions about loss of gases).

This is a transversal study of a cohort of women in reproductive age recruited from May 2016 to June 2018. The clinical and US evaluation were performed at the same medical visit. Patients signed the consent term and answered the questionnaires (King's health quality of life questionnaire, FSF-I (Female Sexual Function - Index, and a scale of anal incontinence) before the ultrasonographic exams. The USG evaluation was performed using GE Voluson 730 expert systems with RAB 8- 4 Mhz volume transducers with an 85-degree acquisition angle. The exams were performed with patient in supine position with hip flexed and using slightly abduced, after voiding. The US transducer was placed on the perineum in the midsagittal position and volumes were obtained at rest, at maximum Valsalva, and perineal contraction. The volumes datasets were analyzed offline by of the authors. They were blinded and the average values were considered.

The studied parameters was the hiatal area (HA), the antero-posterior diameter (PA), transverse diameter (TD) and the muscle thickness (MT). The measures were obtained by the OmniView VCI mode.

Statistical analysis was performed using student t, ANOVA and Tukey. P value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 50
* reproductive age

Exclusion Criteria:

* bad quality of 3D US images
* post- menopause
* vulvovaginitis
* urinary incontinence
* Human papillomavirus vulvar disease (condyloma acuminata)
* previous pelvic floor surgery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Reproductive age women, followed in Family Planning Service and Urogynecology Service of Federal of São Paulo University recruited from May 2016 to June 2018.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
3D US pelvic floor evaluation of transverse diameter of vagina | One day
  Evaluation of transverse diameter of vagina, in cm, by 3D pelvic floor ultrasound

SECONDARY OUTCOMES:
3D US pelvic floor evaluation of thickness of pubovisceral muscle | One day
  Evaluation of thickness of pubovisceral muscle, in cm , by 3D pelvic floor ultrasound
3D US pelvic floor evaluation of Hiatal area | One day
  Evaluation of Hiatal area in cm3, with measures made by 3D pelvic floor ultrasound
Impact of the delivery in quality of life - regarding urinary incontinence | One day
  Evaluation of the impact of delivery in women's quality of life measured by the King's Health Questionnaire score. ( Score range from 0-100, bigger values are associated with worse quality of life)
Impact of the delivery in quality of life - regarding sexual life | One day
  Evaluation of the impact of delivery in women's quality of life measured by FSF-I score ( Score range from 4-99, considered normal over 26)
Impact of the delivery in quality of life - regarding anal incontinente | One day
  Evaluation of the impact of delivery in women's quality of life measured by the score of anal incontinence scale (ocorre range from 0-12, bigger values are associated with worse quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Maria HM Bianchi-Ferraro, PhD, Study Director — Federal University of São Paulo
Locations (1):
- Service of Family Planning ang Urogynecology Service of Department of Gynecology of FEDERAL UNIVERSITY OF SAO PAULO - UNIFESP, São Paulo, São Paulo, Brazil